CLINICAL TRIAL: NCT05916755
Title: Identification of Predictive Biomarkers of Response to Chemotherapy and Immune Checkpoint Inhibitors in Early Triple Negative Breast Cancer: an Integrative Multiomics Platform
Brief Title: Predictive Biomarkers of Response to Checkpoint Inhibitors in Triple Negative Breast Cancer: a Multiomics Platform
Acronym: PORTRAIT
Status: Recruiting | Type: Observational
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)165-2021
Record Dates: First submitted 2023-05-08; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Triple Negative Breast Cancer
Keywords: Circulating biomarkers; clinical tool; immune checkpoint inhibitors; integrative algorithm; microbiome; multiomics; neoadjuvant chemotherapy; predictive biomarkers; radiomics; RNA-Sequencing; triple negative breast cancer; WGS
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Base Sequence; pembrolizumab; Drug Therapy; Carboplatin; taxane; Anthracyclines; Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, Blood samples, Stool, Saliva
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Pembrolizumab + neoadjuvant chemotherapy
  Interventions: Diagnostic Test: Whole Genome Sequencing; Diagnostic Test: RNA-Sequencing; Diagnostic Test: Microbiome analysis; Diagnostic Test: ctDNA analysis; Diagnostic Test: TCR-β repertoire sequencing; Diagnostic Test: PBMCs phenotyping; Drug: Pembrolizumab; Drug: Chemotherapy
- Cohort B: Neoadjuvant chemotherapy
  Interventions: Diagnostic Test: Whole Genome Sequencing; Diagnostic Test: RNA-Sequencing; Diagnostic Test: Microbiome analysis; Diagnostic Test: ctDNA analysis; Diagnostic Test: TCR-β repertoire sequencing; Diagnostic Test: PBMCs phenotyping; Drug: Chemotherapy

INTERVENTIONS:
Diagnostic Test: Whole Genome Sequencing — Whole genome sequencing (WGS) will be performed in tumor tissue from baseline and from residual disease after neoadjuvant chemotherapy (NACT), if present.
  Other Names: WGS
Diagnostic Test: RNA-Sequencing — RNA-Sequencing will be performed in tumor tissue from baseline and from residual disease after NACT (if present).
Diagnostic Test: Microbiome analysis — Microbiome analysis will be performed in stools and saliva before, during NACT and at the end of adjuvant systemic therapy if adjuvant systemic therapy is clinically indicated.
Diagnostic Test: ctDNA analysis — ctDNA analysis will be performed in plasma before and during NACT.
Diagnostic Test: TCR-β repertoire sequencing — TCR-β repertoire sequencing will be performed in plasma before and during NACT.
Diagnostic Test: PBMCs phenotyping — PBMCs phenotyping will be performed in plasma before and during NACT.
Drug: Pembrolizumab — Pembrolizumab will be given in combination with standard NACT.
  Groups: Cohort A
Drug: Chemotherapy — Standard NACT will be given.
  Other Names: Carboplatin, taxane, anthracycline, cyclophosphamide

SUMMARY:
Patients with stage II-III Triple negative breast cancer (TNBC) candidates to receive neoadjuvant chemotherapy (NACT) +/- immune checkpoint inhibitor (ICI) will be included. Several samples from different tissues will be analyzed through different omics to establish predictive biomarkers of response to the treatment. Multiple algorithms will then be used to look for an integrative predictive algorithm that incorporates multi-parameter inputs in order to develop a clinical tool to assist clinicians in the process of treatment decision-making in TNBC.

DETAILED DESCRIPTION:
The combination of pembrolizumab, an immune checkpoint inhibitor (ICI), with neoadjuvant chemotherapy (NACT) increases pathologic complete response (pCR) and event-free survival (EFS) in patients with early triple negative breast cancer (eTNBC). However, not all patients equally benefit from a treatment that may have relevant adverse events (AEs).

Objectives: (1) To establish predictive biomarkers of response to NACT + ICI in eTNBC by correlating data coming from different layers of omics performed in different tissues, together with imaging, with pCR, EFS, and overall survival (OS). (2) To integrate data generated from (1), and clinical data, and explore multivariate predictive models of response to NACT + ICI.

Methods: Patients with stage II-III TNBC candidates to receive NACT +/- ICI will be included. Collected samples and type of analysis: (1) Tumor tissue (baseline and from residual disease after NACT): whole genome sequencing (WGS) and RNA-Seq will be performed (Hartwig sequencing platform and analytical pipeline), tissue immune phenotyping (PD-L1, T and B infiltrating lymphocytes, among others), and microbiome analysis (16S rRNA); (2) Blood (before and during NACT): circulating tumor DNA (ctDNA) analysis (targeted gene panel and shallow WGS), T-cell receptor beta (TCR-β) repertoire sequencing and analysis (ImmunoSeq hsTCRβ kit and immunoSEQ), and peripheral blood mononuclear cells (PBMCs) phenotyping; (3) Stools and saliva (before and during NACT): microbiome analysis (16S rRNA); (4) Breast MRI imaging (before and after NACT): radiomics analysis. Multiple algorithms including Multiple Kernel Learning, Multi-Omics Factor Analysis (MOFA) and Method for the Functional Integration of Spatial and Temporal Omics data (MEFISTO) will then be used to look for an integrative predictive algorithm that incorporates multi-parameter inputs. The aim is to provide more personalized treatment efficacy and risk for relapse estimates.

Expected outcome: To develop a clinical tool to assist clinicians in the process of treatment decision-making in eTNBC, in order to maximize patient's benefit and quality of life, while minimizing AEs and financial burden to the health system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented TNBC (negative human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PgR] status)
* Stage 2 - 3 defined by the American Joint Committee of Cancer (AJCC) staging criteria 8th edition for breast cancer as assessed by the investigator based on radiological and/or clinical assessment
* Patient is a candidate to receive NACT with or without ICI as assessed by the investigator
* Patient is ≥ 18 years old at the time of consent to participate in this trial

Exclusion Criteria:

* Metastatic disease on imaging (stage 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II-III TNBC candidates to receive NACT +/- ICI will be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate at definitive surgery | after neoadjuvant treatment and surgery, up to approximately 27-30 weeks
  The rate (given as a percentage) of patients with a pCR at definitive surgery using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) from the American Joint Committee on Cancer (AJCC) staging criteria
Event-free survival (EFS) | Up to approximately 60 months
  EFS is defined as the time from the start of neoadjuvant treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause
Overall survival (OS) | Up to approximately 60 months
  OS is defined as the time from starting neoadjuvant treatment until death due to any cause
Identification of biomarkers to predict clinical outcomes (pCR at definitive surgery, EFS, OS). | After all data are analyzed, up to approximately 60 months
  The clinical data (pCR at definitive surgery, EFS, OS) will be integrated with the results from the multiomics platform and multivariate predictive models of response to neoadjuvant chemotherapy (NACT) + immune checkpoint inhibitor (ICI) will be explored. Precisely, the multiomics platform will analyze:
  1. RNA-Sequencing of the initial tumor and residual disease (if present)
  2. microbiome analysis of the saliva and feces,
  3. circulating tumor DNA (ctDNA) analysis (targeted gene panel and shallow WGS),
  4. Tissue immune phenotyping,
  5. T-cell receptor beta (TCR-β) repertoire sequencing and analysis using ImmunoSeq hsTCRβ kit and immunoSEQ,
  6. Breast MRI imaging (before and after NACT),
  Multiple algorithms including Multiple Kernel Learning, Multi-Omics Factor Analysis (MOFA) and Method for the Functional Integration of Spatial and Temporal Omics data (MEFISTO) will then be used to look for an integrative predictive algorithm that incorporates multi-parameter inputs.

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided